CLINICAL TRIAL: NCT02327780
Title: The Effectivness of FODMAP Diet in Israel in Relieving Symptoms of Patients With Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 407-14-TLV
Record Dates: First submitted 2014-12-24; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

ARMS (1):
- FODMAP diet (Other): participants will be put on a low FODMAP diet.
  Interventions: Other: FODMAP diet

INTERVENTIONS:
Other: FODMAP diet

SUMMARY:
Treatment of IBS is very problematic. Despite the wide range of pharmacological and non-pharmacological therapies, there is no universally accepted approach. In recent years, the low FODMAP diet has been developed, a dietary approach that aims to relieve the symptoms of IBS. FODMAPs (Fermentable Oligosaccharides, Di-saccharides, Mono-saccharides and Polyols) are a group of dietary sugars that may be poorly absorbed in the small intestine and fermented by bacteria to produce gas. Ingestion of FODMAPs may also result in alterations in fluid content in the colon and trigger functional gut symptoms in some individuals. This study aims to examine the effectiveness of the FODMAP diet in Israel in improving symptoms of IBS compared to the standard dietary advice.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfillment of the Rome III criteria for IBS.
2. Aged 18-77 years at the time of screening.
3. Provision of written informed consent.
4. Commitment of availability throughout the 10 week study period.
5. Availability of at least one GI imaging study during the last 5 years (colonoscopy, sigmoidosopy, abdominal ultrasonography, barium enema) for subjects older than 50 years.

Exclusion Criteria:

1. Major abdominal surgery in the past.
2. The presence of any active (organic) GI disease.
3. Past or present major medical or psychiatric illness.
4. Any concomitant disease.
5. Alarming symptoms (rectal bleeding, weight loss, etc.)
6. Pregnancy.
7. Family history of colorectal carcinoma or IBD, under the age of 50.
8. Abnormal laboratory studies (blood biochemistry, liver enzymes, complete blood count), abnormal thyroid function.
9. Non-adjusted diet in the case of lactose or gluten intolerance.
10. Recent travel to regions with endemic parasitic diseases.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome (IBS) severity score | 9 weeks
IBS quality of life score | 9 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Unit, Sourasky Medical Center, Tel Aviv, Israel